CLINICAL TRIAL: NCT00840255
Title: Treatment of Insomnia in Military Veterans:Phase 2
Brief Title: Brief Behavioral Treatment of Insomnia in Military Veterans: Phase 2 (BBTIMVII)
Acronym: BBTIMVII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anne Germain, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO08070327; NIMH: 1 R34 MH080696
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Insomnia
Keywords: Chronic Insomnia lasting more than 1 month
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breif Behavioral Treatment of Insomnia (Active Comparator): Effective behavioral insomnia treatments are typically delivered over an 8-week period. This format may not be easily exportable to primary and community care settings where military returnees and veterans seek help. The goal here is to test the effects of a 4-week behavioral treatment that targets chronic insomnia (lasting >1 month) in service members returning from Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF), and who present with the typical psychiatric comorbidities associated of combat-related anxiety and mood disorders and stress reactions.
  Interventions: Behavioral: BBTI-MV
- Information Control (Other): This arm of the study does not receive the Brief Behavioral Treatment for Insomnia. This arm will act as the control arm.
  Interventions: Other: Information Control

INTERVENTIONS:
Behavioral: BBTI-MV — Twenty participants will be randomized to BBTI-MV. As previously described, the intervention will be delivered over 4 consecutive weeks, which include individual face-to-face visits on Weeks 1 and 3, and telephone appointments on Weeks 2 and 4. Interventions will be delivered at Western Psychiatric Institutes and Clinic. If possible, (according to space availability), the face-to-face sessions may also be conducted at the VAPHS clinics or at Reserve and Veterans Centers locally and regionally to strengthen our relations with local care and services providers and centers, and to facilitate future collaborative efforts. The duration of the first treatment visit is 45-minutes, and the follow-up visit on Week 3 will last no more than 30 minutes. Brief (<20 minutes) telephone sessions will be conducted on Weeks 2 and 4.
  Arms: Breif Behavioral Treatment of Insomnia
Other: Information Control — Participants will receive two brochures from the American Academy on Sleep Medicine of Sleep Hygiene and on Insomnia. The therapists will read the content of the 2 brochures with participants, and discuss how the information provide relates to individual participants' sleep experiences. No recommendations for altering sleep schedules will be made by the assigned therapist. Participants will be instructed to read these two brochures over the course of the following week, and to consider how the information provided in the brochures related to their own sleep patterns
  Arms: Information Control

SUMMARY:
The purpose of this study is to adapt and test the effects of a 4-week behavioral treatment that targets chronic insomnia (lasting >1 month) in service members returning from Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF), finalizing a treatment manual.

DETAILED DESCRIPTION:
Insomnia is one of the most common reasons for referral to mental health services in active duty personnel. Chronic insomnia often persists post-deployment, contributes to poor mental and physical health outcomes, and requires targeted interventions. Effective behavioral treatments of insomnia have not been adapted and tested for the treatment of chronic insomnia comorbid to combat-related mental disorders and stress reactions. In addition, effective behavioral insomnia treatments are typically delivered over an 8-week period. This format may not be easily exportable to primary and community care settings where military returnees and veterans seek help. The goal is to adapt and test the effects of a 4-week behavioral treatment that targets chronic insomnia (lasting >1 month) in service members returning from Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF), and who present with the typical psychiatric comorbidities associated of combat-related anxiety and mood disorders and stress reactions. We call this intervention the Brief Behavioral Treatment of Insomnia for Military Veterans (BBTI-MV). The proposed study includes two phases. The specific aims of Phase II are: (1) To explore the effects of BBTI-MV on sleep and daytime symptoms of psychiatric distress. We anticipate that participants randomized to BBTI-MV will show a higher categorical response rate and remission for sleep symptoms than subjects randomized to IC. (2) To evaluate in a preliminary manner the durability of therapeutic gains and by conducting a naturalistic follow-up assessment six months post-treatment in responders. (3) To explore whether the nature of combat-related experiences, time since deployment and since, return to the US, deployment theater, medication use and change in dosage, mood and anxiety or disorders affect sleep treatment adherence and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18 years old and older
2. Military returnees from OIF/OEF
3. Meet diagnostic criteria for chronic insomnia as defined by:

   a. Complaint of sleep latency >30 minutes, or wake time after sleep onset >30 minutes, or Sleep Efficiency <85%, or a complaint of non-restorative sleep
   * Frequency of insomnia complaint >3 times per week;
   * Duration of insomnia complaint >1 month
   * Associated with at least one daytime consequences
4. If using sleep medications, medication and dosage have not been changed in the past month, and will remain unchanged for the duration of the acute treatment phase of the study (i.e., 4 weeks)
5. If using other psychotropic medications, medication and dosage have not been changed in the past 2 months, and will remain unchanged for the duration of the acute treatment phase of the study (i.e., 4 weeks)

Exclusion Criteria:

1. Active duty personnel, or reservists/national guards scheduled to re-deploy if their departure date is < 2 months from the consent date
2. Untreated, current, and severe PTSD as determined on the SCID.
3. Untreated, current, and severe Major Depressive Disorder as determined by the Structured Clinical Interview for DSM-IV and a score > 30 on the Beck Depression Inventory
4. Psychotic or bipolar disorder
5. Current substance or alcohol use disorder as determined by the SCID or by positive drug toxicology results
6. Unstable medical condition
7. Hospitalization in the previous 2 weeks for a medical condition or surgery for which recovery overlaps with the study onset and duration
8. Seizure disorder or open skull brain injury.
9. Current sleep disorders such as nightmare disorder, restless legs syndrome, or suspected sleep disorder requiring polysomnographic assessment, such as obstructive sleep apnea or periodic leg movements.
10. Sleep apnea revealed during the screening sleep study.
11. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Diary | Weekly
Pittsburgh Sleep Quality Index (PSQI) | Baseline and Post Intervention
PSQI Addendum for PTSD (PSQIA) | Baseline and Post
Sleep Quality defined by: PIRS-20 and ISI | Screening,Baseline, and Post

SECONDARY OUTCOMES:
PTSD symptom severity as measured by the CAPS | Screening
Depression: BDI | Baseline and Post
Anxiety: BAI | Baseline and Post
Medical History: MHQ, MEDHIST_2WK, MOS | Screening, Baseline, and Post
Trauma History: THQ,CES,PCL-C,ICG | Screening, Baseline, and Post
Post Sleep Self Report: PSEQ-SV and POST | Screening
Sleepiness: EPWORTH, BASS | Screening, Baseline, and Post
Mood and Behavior: BIS/BAS, SMITH, PANAS | Screening, Baseline, and Post
Expectations and Satisfaction: TEQ-94, Client Satisfaction Survey | Baseline and Post

CONTACTS AND LOCATIONS:
Overall Officials: Anne Germain, PhD, Principal Investigator — University of Pittsburgh, Department of Psychiatry
Locations (1):
- Western Psychiatric Institute & Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Germain A, Richardson R, Stocker R, Mammen O, Hall M, Bramoweth AD, Begley A, Rode N, Frank E, Haas G, Buysse DJ. Treatment for insomnia in combat-exposed OEF/OIF/OND military veterans: preliminary randomized controlled trial. Behav Res Ther. 2014 Oct;61:78-88. doi: 10.1016/j.brat.2014.07.016. Epub 2014 Aug 12. PMID 25194223